CLINICAL TRIAL: NCT01252095
Title: An Open-label, Single Centre Phase I Study of the Safety and Tolerability of PG545 in Patients With Advanced Solid Tumours
Brief Title: Study of the Safety and Tolerability of PG545 in Patients With Advanced Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unexpected injection site reactions.
Sponsor: Zucero Pty Ltd (Industry)
Collaborators: Statistical Revelations Pty Ltd (Unknown); Datapharm Australia Pty Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PG545101
Record Dates: First submitted 2010-11-30; First posted 2010-12-02 (Estimated); Results first posted 2012-08-02 (Estimated); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Advanced Solid Tumours
Keywords: PG545; Phase I; Progen; antimetastatic; antiangiogenic; advanced cancer patients; solid tumors; solid tumours

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PG545 (Experimental)
  Interventions: Drug: PG545

INTERVENTIONS:
Drug: PG545 — PG545 Lyophilized Powder for Subcutaneous Injection. Patients will be dosed once weekly until they exhibit disease progression, are discontinued for reasons of tolerability, or the study reaches its defined end-point. This study is a dose escalation study with doses of 25 mg to 500 mg planned.

SUMMARY:
This first-in-human study aims to establish the maximum tolerated dose of PG545 and to evaluate its safety in subjects with advanced solid tumours. In addition the study will explore whether PG545 exposure results in changes to chemicals produced by the body that are associated with cancer growth and spread.

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Histological or cytological documentation of non hematologic, malignant solid tumour.
* Have failed at least one previous therapeutic regimen.
* Measurable disease according to RECIST 1.1.
* Life expectancy >= 12 weeks
* ECOG Performance Status of 0 or 1
* Written, signed and dated informed consent
* Able and willing to meet all protocol-required treatments, investigations and visits.
* Have adequate organ function

Exclusion Criteria:

* Clinically significant non-malignant disease.
* Active CNS metastases.
* Subjects with uncontrolled diabetes.
* History of clinically significant adverse drug reaction to heparin or other anti-coagulant agents
* History of immune-mediated thrombocytopaenia or other platelet abnormalities or other hereditary or acquired coagulopathies.
* Concomitant use of aspirin (> 150 mg/day), NSAIDs (except COX-2 selective inhibitors), vitamin K antagonists (other than low-dose prophylactic use), heparin within two weeks prior to randomisation, or other anti-platelet drugs.
* History of severe allergic, anaphylactic or other significant adverse reaction to radiographic contrast media
* Known seropositivity to the human immunodeficiency virus (HIV)
* Women who are pregnant or breast-feeding.
* Women of child-bearing potential and male subjects who are partners of women of childbearing potential who are unable or unwilling to practice a highly effective means of contraception.
* Active substance abuse
* Subjects who have received an investigational agent within 28 days prior to Cycle 1 Day 1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Millward, MBBS, Principal Investigator — Head of Department, Medical Oncology, Sir Charles Gairdner Hospital
Locations (1):
- Linear Clinical Research Ltd, Nedlands, Western Australia, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from Perth oncology clinics and treated under the PG545101 protocol at the dedicated phase I unit, Linear Clinical Research Ltd. The recruitment period was November 2010 to October 2011.
Groups:
- 25 mg Dose: 25 mg PG545/week
- 50 mg Dose: 50 mg PG545/week
Period: Overall Study
Arm/Group | 25 mg Dose | 50 mg Dose
Started | 3 | 1
Completed | 2 | 1
Not Completed | 1 | 0
Not completed — Disease progression | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg Dose | 50 mg Dose | Total
Number analyzed (Participants) | 3 | 1 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (5) | 57 | 62 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Australia | 3 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) Based on DLT
Description: The primary objective of this study is the determination of the MTD. Due to the premature termination of the study the MTD could not be determined. The outcome measure presented is the number of DLTs per cohort.
Time Frame: Following first 1 month cycle
Population: Patients had to complete cycle 1 per protocol.
Measure: Number; unit: DLTs
Arm/Group | 25 mg Dose | 50 mg Dose
Number analyzed (Participants) | 2 | 1
DLTs | 0 | 1

ADVERSE EVENTS:
Time Frame: Patients were on treatment for up to 51 days. Adverse events were collected from signing of informed consent.
Arm/Group | 25 mg Dose | 50 mg Dose
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/1
Other Adverse Events (participants affected / at risk) | 3/3 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 25 mg Dose (N=3) | 50 mg Dose (N=1)
Redness at injection site (Skin and subcutaneous tissue disorders) | 1 (4) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 3 (14) | 0 (0)
Cellulitus around umbilicus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Facial flushing (Vascular disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (2)
Local reactions (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)

LIMITATIONS AND CAVEATS:
Early termination due to unexpected injection site reactions leading to small numbers of subjects analyzed. An MTD could not be determined for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No data may be published or presented from the study except with the prior written consent of Progen. Progen reserves the right to a 30-day review and approval of all manuscripts related to the study prior to publication.